CLINICAL TRIAL: NCT06818565
Title: Comparison of Efficacy and Safety of Ceftazidime Avibactam Versus Extended Infusions of High Dose Meropenem in Patients of ACLF With Nosocomial Infections.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-20
Record Dates: First submitted 2025-02-01; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Meropenem; avibactam, ceftazidime drug combination; Teicoplanin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meropenem (Active Comparator): Meropenem 2gm TDS over 3 hours infusion Teicoplanin 400 mg iv BD for 3 doses f/b 400 mg iv OD
  Interventions: Drug: Meropenem Injection; Drug: Teicoplanin
- Ceftazidime avibactam (Experimental): Ceftazidime avibactam 2.5 gm iv TDS. Teicoplanin 400 mg iv BD for 3 doses f/b 400 mg iv OD
  Interventions: Drug: Ceftazidime-avibactam; Drug: Teicoplanin

INTERVENTIONS:
Drug: Meropenem Injection — Meropenem 2 gm iv TDS
  Arms: Meropenem
Drug: Ceftazidime-avibactam — Ceftazidime-avibactam 2.5 gm iv TDS
  Arms: Ceftazidime avibactam
Drug: Teicoplanin — Teicoplanin 400 mg iv BD 3 doses followed by 400mg iv OD

SUMMARY:
Acute on chronic liver failure patients are at high risk for nosocomial infections due to liver dysfunction, which impairs immune responses and increases vulnerability to infections. Key factors contributing to nosocomial infections in ACLF patients include ascites, use of invasive devices, and recent hospitalization, frequent need for broad spectrum antibiotics. Multidrug resistance is a growing issue, making treatment more challenging, common pathogens involved are gram negative bacteria such as Escherichia Coli and Klebsiella pneumoniae. Surveillance data show increasing carbapenem resistant enterobacterales (CRE) infection rates in cirrhotics, with high morbidity and mortality rates. The impact of these nosocomial infections is profound, significantly worsen outcomes in ACLF patients, leading to prolonged hospitalizations, increased health care costs and higher mortality rates. Early detection and effective antibiotic stewardship are essential to manage antibiotic resistance and improve patient outcomes. In this study we aim to compare efficacy and safety of Ceftazidime avibactam versus extended infusions of high dose Meropenem in patients of ACLF with nosocomial infections.

DETAILED DESCRIPTION:
Hypothesis - We hypothesize that ceftazidime-avibactum would be superior and an effective carbapenem sparing agent compared to extended high dose carbapenems as empirical therapy in management of nosocomial infections caused by carbapenem resistant organisms in patients with ACLF.

Aim -To compare the efficacy and safety of Ceftazidime avibactam and extended infusions of high dose Meropenem as emperical antibiotic in patients of ACLF with nosocomial infections caused by carbapenem resistant organisms.

Primary objective:

• To compare the efficacy of Ceftazidime avibactam over extended infusions of high dose carabapenem as emperical antibiotic in achieving clinical response at day 3 in patients of ACLF with suspected nosocomial infections.

Secondary objectives:

* To study the spectrum of nosocomial infections, bacterial DNA and resistance genes in the context of nosocomial infections in ACLF
* Proportion of patients requiring escalation/de-escalation of antibiotics at day 3
* Incidence of clinical and microbiologic response at day 5 and day 7
* Time to escalation of antibiotics in both groups
* Transfer to icu, mortality, and progression of organ failures and worsening of AARC scores by grade I, SOFA score by point 2.
* Microbiologic outcome (Eradication/Persistence)
* To identify biomarkers of host response to empirical antibiotic regimen
* Transplant free survival at day 15 and day 28
* Proportion of patients made eligible for transplant day 7. A prospective, Randomized Control Trial. Single centre, Open label, Block randomization will be done, it will be implemented by IWRS method. This study will be conducted in Department of Hepatology, ILBS.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. ACLF as per APASL criteria
3. ACLF patients with nosocomial infections caused by carbapenem resistant organism (defined as suspected or documented evidence of infection after 48 hours of hospitalization) requiring antibiotics.

Exclusion Criteria:

1. Severe septic shock with MOF requiring escalation of antibiotics
2. Patients having known allergies to meropenem or Ceftazidime Avibactam
3. Culture sensitivity showing isolate non susceptible to study drug being investigated.
4. Already on either regimen, receiving meropenem or Ceftazidime Avibactam >48 hours.
5. On mechanical ventilator support PF ratio < 300.
6. Patients on immunosuppression medication
7. HCC or other malignancies
8. CKD
9. CAD
10. Pregnancy or Lactation
11. Post Liver Transplantation
12. Refusal to consent
13. PLWHA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of ACLF patients with nosocomial infection by carbapenem resistant organisms showing clinical response at the end of treatment. | Day 3

SECONDARY OUTCOMES:
Time to escalation or descalation of antibiotics | within 3 days
Progression in terms of organ dysfunction/failure at day 5 and 7. | day 5 and 7
Incidence of adverse events in both groups. | within 7 to 10 days
Duration of hospital and ICU stay | day 28
Mortality at day 15 and day 28 | day 15 & 28

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided